CLINICAL TRIAL: NCT06974682
Title: Effect of Target Temperature Management on Intestinal Flora and Its Metabolites in Patients With Cardiac Arrest
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Tang Ziren, professor, Capital Medical University
Other Study IDs: 2025-4-10-8
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Arrest (CA)
Keywords: Cardiac Arrest; intestinal flora; Intestinal metabolites; Macrogenome
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the self-control design, this study explored the dynamic regulation of target temperature management therapy (TTM) on intestinal flora structure and metabolites of patients after cardiopulmonary resuscitation (CPR). This study is a single-center prospective observational study. Patients with spontaneous circulation recovery (ROSC) after CPR and TTM were included before and after self-hypothermia treatment, and the time series changes of intestinal flora and metabolites at some representative time points before and after treatment were compared. Thirty-five adult patients (age ≥18 years) who met the admission criteria were included. Before TTM treatment (0h after ROSC, baseline), 48 h after TTM warming (T1) and 48 h after rewarming (T2), fecal samples (macro-gene sequencing) and blood samples (metabonomics) were collected to analyze the changes of intestinal flora and metabolites in patients with cardiac arrest, and to screen the differential flora and metabolites regulated by TTM and their dynamic correlation.

ELIGIBILITY:
Inclusion Criteria:

* (1).18 years old and above; (2) Successful resuscitation after cardiopulmonary resuscitation (including chest compressions, electric shock defibrillation, etc.) and target temperature management;

Exclusion Criteria:

* (1) Pregnant or lactating women; (2) Patients with intestinal dysfunction: including severe acute intestinal injury, intestinal obstruction or other diseases that affect the normal function of the intestine; (3) Immunosuppression status: such as patients who use immunosuppressants, or patients with obvious immune dysfunction (such as HIV infection, organ transplant patients, etc.); (4) Those who have recently undergone intestinal surgery or endoscopy; (5) The patient or his family failed to sign the informed consent or refused to participate in the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successful cardiopulmonary resuscitation (CPR) were transferred to the emergency intensive care unit for further standardized management.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal flora structure | one year
  Diversity of intestinal flora

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chaoyang hospital, Beijing, Beijing 100020, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors